CLINICAL TRIAL: NCT04147793
Title: Case Control Study to Investigate the Use of Urethral Pressure Profile Measurement in Children
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 269193
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Dysfunctional Voiding; Stress Incontinence, Urinary
Keywords: child; Adolescent; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Controls: patients attneding for surgery with no known bladder disease
- Overactice sphincter: those with evidence of dysfunctional voiding
- Underactive sphincter: those with genuine stress incontinence

SUMMARY:
The bladder has a muscle that acts like a tap called the sphincter. Just like a tap, when pee is stored the sphincter muscle is closed and during peeing the sphincter opens. Sometimes the sphincter tap does not work properly and can cause problems. If the sphincter is weak there can be urine leak (incontinence). If the sphincter is too strong bladder might not empty properly.

Children who require investigation of their urinary problems are usually assessed with non-invasive tests. Sometimes investigation is with a more invasive test videourodynamics or video cystometrogram (VCMG; this test requires the insertion of catheters into the bladder and rectum. This test provides only indirect information about sphincter function.

It would be helpful to have a more direct test of the sphincter. It will allow better targeted treatments of sphincter problems which are often therapeutically challenging. Urethral pressure profile is a test used in adults to assess the sphincter. Although it has been described in children normal values have not been described.

The research project is to define urethral pressure profile values in children and young people with normal, weak and overactive sphincters.

Urethral pressure profile measurement is invasive as it requires the insertion of a special catheter. It will therefore be performed at the time of other invasive procedures eg VCMG or urology surgery under general anaesthetic.

The study will be conducted at single site, which is a children's hospital. The study will be an observational case controlled study with three arms: controls, those with overactive sphincters and those with underactive sphincters. The study is intended to run over three years.

DETAILED DESCRIPTION:
Rationale Bladder problems in children are common resulting in incontinence and social distress.

The bladder performs two functions: storage and emptying. It has two components that act synchronously with each other and allow it to achieve this: the detrusor and the sphincter complex. The detrusor is the muscle in the wall of the bladder. The sphincter complex is a group of muscles that act on the urethra, which is the outlet of the bladder. During storage the detrusor muscle is relaxed while the sphincter complex is closed. During bladder emptying the detrusor muscle contracts while the sphincter relaxes. Abnormal function of either component will result in abnormal bladder function including lower urinary tract symptoms (including frequency urgency, incontinence, difficulty voiding) and danger to the kidneys. Specifically, abnormality of the sphincter will result in either incontinence during storage, or obstructive problems during voiding.

Establishing a bladder diagnosis in children is helped by performing a test of bladder function. In the majority of children this can be done with non-invasive assessments that include bladder diary, flow rates, flow patterns residual volume measurements and electromyogram (EMG) using skin electrodes. However, in some children non-invasive testing is not able to provide enough information and so videocystometry (VCMG), or urodynamics, are performed. These are more invasive tests. Catheters are inserted into the bladder and abdomen (usually the rectum) to measure pressures generated by the detrusor. The flow rate is measured during emptying. Combining this with x-ray fluoroscopy provides additional anatomical information. VCMG provides direct information about the detrusor. Standard VCMG in children do not currently provide direct information about the tone of the sphincter. Information about sphincter function is provided indirectly by measuring the pressures during leaking, or during voiding from analysis of flow, pressure and X-ray imaging.

The investigators believe that there is a need to develop a direct diagnostic test of sphincter function in children. The investigators have a practice where children are seen with both sphincter underactivity and overactivity. Sphincter under- activity is most commonly seen in children with abnormal bladder function as a result of neurological disease (neuropathic bladder). Sphincter incompetence can be difficult to treat in children . A diagnostic test that can better define the condition may allow better targeted treatments. Sphincter overactivity will result in a poorly emptying bladder. However poor bladder emptying can also result from detrusor underactivity. In patients with incomplete bladder emptying it can be difficult to distinguish whether the condition is as a result of underactive detrusor or overactive sphincter (e.g. dysfunctional voiding or high-tone non-relaxing sphincter type conditions). The distinction is important because the two conditions require very different treatments.

There are tests of sphincter function:

* Abdominal leak point pressure (ALPP). This is performed during VCMG. It is the lowest pressure measured in the bladder at which leaking happens during a series of increasingly more forceful Valsalva manoeuvres or cough. It is dependent on incontinence occurring. It is an indirect test of sphincter function; the pressure in the bladder at the precise moment of leaking provides the measure of sphincter tone. It can sometimes be difficult to get children to perform this test.
* Retrograde leak point pressure (RLPP). This is a test of sphincter weakness performed in men. A catheter is inserted into the male urethra and x-ray contrast is injected. The RLPP is the lowest pressure required for the contrast to overcome the sphincter and enter the bladder. The test requires an adequate length of urethra and so can only practically be used in males.
* Electromyogram (EMG). Electrodes can be used to measure electrical activity. In children skin electrodes are used; this makes it difficult to distinguish between pelvic floor and sphincter activity. Invasive needle electrodes can be used to specifically target the sphincter, but this is cumbersome, invasive and offered in very few units. EMG provides qualitative information on whether there is overactivity of muscles being recorded.
* Videocytometogram (VCMG). Described above, this can give an assessment of the presence of overactive sphincter during voiding based on an evaluation and opinion from pressure flow and x-ray appearance during voiding.
* Urethral pressure profile (UPP). Pressure recording catheters are passed through the sphincter to directly measure the pressure applied by the sphincter. This technique can be used to identify both overactive and underactive sphincter activity. The technique of UPP is used to derive the maximum urethral closure pressure (MUCP). This is the maximum difference between the urethral pressure and the intravesical pressure .

Urethral pressure profile measurement carries great promise as a diagnostic test. It has been validated in adults to diagnose sphincter weakness as well as diagnosing high tone non-relaxing sphincter disorders. The test is easy to perform. Its use has previously been described in children; in this early description it was found not to be helpful in diagnosing bladder outlet obstruction. However, one of the conditions for which UPP shows promise is high tone non-relaxing sphincter, which was not described as a clinical entity until a later time. However UPP has not been validated in children.

The investigators propose a study to investigate the use of UPP in children. The hypothesis is that there are values and characteristics of the UPP that can distinguish control patients from those with either sphincter underactivity and sphincter overactivity.

The investigators will measure MUCP in three patient groups and compare the values. These three groups will be discussed in more detail:

Controls. These patients will have no known bladder disease. This will be asked in pre-recruitment checks. The patients will complete a validated questionnaire- the Dysfunctional Voiding Scoring System (DVSS). A normal score, ie less than less than 6 in girls and less than 9 in boys, will indicate that the child has no significant urinary symptoms.

Measurement of UPP is invasive, requiring a fine catheter to be passed through the urethra; performing it in an otherwise well child presents difficulties. UPP's will therefore be measured under general anaesthetic in children who require general anaesthesia for other urological conditions, eg renal stones. Such a child will have much larger instruments passed through the urethra as part of their urology surgery so that performing a urethral pressure profile should not significantly add to their discomfort or risk. General anaesthetic will be induced with an inhalational anaesthetic agent. A light level of general anaesthesia will then be maintained with the same inhalation agent. This will avoid administration of intravenous anaesthetic agents which may affect UPP values . A light inhalational general anaesthesia has not been shown to affect UPP measurements. After the UPP measurement has been performed, which is expected to take less than five minutes, general anaesthesia will then be changed to a level sufficient for the planned urological procedure.

Overactive sphincter These patients have presented to the bladder service with problems because of abnormality of sphincter activity. These children will be expected to have high tone sphincters. They may have varieties of diagnoses which include high tone non-relaxing sphincter, Fowler's syndrome and dysfunctional voiding. They will commonly have voiding symptoms such as hesitancy, straining, poor stream or the sensation of incomplete emptying. There is, perhaps, surprisingly high incidence of storage symptoms such as frequency urgency and incontinence.

Detailed Description: Rationale Bladder problems in children are common resulting in incontinence and social distress.

The bladder performs two functions: storage and emptying. It has two components that act synchronously with each other and allow it to achieve this: the detrusor and the sphincter complex. The detrusor is the muscle in the wall of the bladder. The sphincter complex is a group of muscles that act on the urethra, which is the outlet of the bladder. During storage the detrusor muscle is relaxed while the sphincter complex is closed. During bladder emptying the detrusor muscle contracts while the sphincter relaxes. Abnormal function of either component will result in abnormal bladder function including lower urinary tract symptoms (including frequency urgency, incontinence, difficulty voiding) and danger to the kidneys. Specifically, abnormality of the sphincter will result in either incontinence during storage, or obstructive problems during voiding.

Establishing a bladder diagnosis in children is helped by performing a test of bladder function. In the majority of children this can be done with non-invasive assessments that include bladder diary, flow rates, flow patterns residual volume measurements and electromyogram (EMG) using skin electrodes. However, in some children non-invasive testing is not able to provide enough information and so videocystometry (VCMG), or urodynamics, are performed. These are more invasive tests. Catheters are inserted into the bladder and abdomen (usually the rectum) to measure pressures generated by the detrusor. The flow rate is measured during emptying. Combining this with x-ray fluoroscopy provides additional anatomical information. VCMG provides direct information about the detrusor. Standard VCMG in children do not currently provide direct information about the tone of the sphincter. Information about sphincter function is provided indirectly by measuring the pressures during leaking, or during voiding from analysis of flow, pressure and X-ray imaging.

The investigators believe that there is a need to develop a direct diagnostic test of sphincter function in children. The investigators have a practice where children are seen with both sphincter underactivity and overactivity. Sphincter under- activity is most commonly seen in children with abnormal bladder function as a result of neurological disease (neuropathic bladder). Sphincter incompetence can be difficult to treat in children . A diagnostic test that can better define the condition may allow better targeted treatments. Sphincter overactivity will result in a poorly emptying bladder. However poor bladder emptying can also result from detrusor underactivity. In patients with incomplete bladder emptying it can be difficult to distinguish whether the condition is as a result of underactive detrusor or overactive sphincter (e.g. dysfunctional voiding or high-tone non-relaxing sphincter type conditions). The distinction is important because the two conditions require very different treatments.

There are tests of sphincter function:

* Abdominal leak point pressure (ALPP). This is performed during VCMG. It is the lowest pressure measured in the bladder at which leaking happens during a series of increasingly more forceful Valsalva manoeuvres or cough. It is dependent on incontinence occurring. It is an indirect test of sphincter function; the pressure in the bladder at the precise moment of leaking provides the measure of sphincter tone. It can sometimes be difficult to get children to perform this test.
* Retrograde leak point pressure (RLPP). This is a test of sphincter weakness performed in men. A catheter is inserted into the male urethra and x-ray contrast is injected. The RLPP is the lowest pressure required for the contrast to overcome the sphincter and enter the bladder. The test requires an adequate length of urethra and so can only practically be used in males.
* Electromyogram (EMG). Electrodes can be used to measure electrical activity. In children skin electrodes are used; this makes it difficult to distinguish between pelvic floor and sphincter activity. Invasive needle electrodes can be used to specifically target the sphincter, but this is cumbersome, invasive and offered in very few units. EMG provides qualitative information on whether there is overactivity of muscles being recorded.
* Videocytometogram (VCMG). Described above, this can give an assessment of the presence of overactive sphincter during voiding based on an evaluation and opinion from pressure flow and x-ray appearance during voiding.
* Urethral pressure profile (UPP). Pressure recording catheters are passed through the sphincter to directly measure the pressure applied by the sphincter. This technique can be used to identify both overactive and underactive sphincter activity. The technique of UPP is used to derive the maximum urethral closure pressure (MUCP). This is the maximum difference between the urethral pressure and the intravesical pressure .

Urethral pressure profile measurement carries great promise as a diagnostic test. It has been validated in adults to diagnose sphincter weakness as well as diagnosing high tone non-relaxing sphincter disorders. The test is easy to perform. Its use has previously been described in children; in this early description it was found not to be helpful in diagnosing bladder outlet obstruction. However, one of the conditions for which UPP shows promise is high tone non-relaxing sphincter, which was not described as a clinical entity until a later time. However UPP has not been validated in children.

The investigators propose a study to investigate the use of UPP in children. The hypothesis is that there are values and characteristics of the UPP that can distinguish control patients from those with either sphincter underactivity and sphincter overactivity.

The investigators will measure MUCP in three patient groups and compare the values. These three groups will be discussed in more detail:

Controls. These patients will have no known bladder disease. This will be asked in pre-recruitment checks. The patients will complete a validated questionnaire- the Dysfunctional Voiding Scoring System (DVSS). A normal score, ie less than less than 6 in girls and less than 9 in boys, will indicate that the child has no significant urinary symptoms.

Measurement of UPP is invasive, requiring a fine catheter to be passed through the urethra; performing it in an otherwise well child presents difficulties. UPP's will therefore be measured under general anaesthetic in children who require general anaesthesia for other urological conditions, eg renal stones. Such a child will have much larger instruments passed through the urethra as part of their urology surgery so that performing a urethral pressure profile should not significantly add to their discomfort or risk. General anaesthetic will be induced with an inhalational anaesthetic agent. A light level of general anaesthesia will then be maintained with the same inhalation agent. This will avoid administration of intravenous anaesthetic agents which may affect UPP values . A light inhalational general anaesthesia has not been shown to affect UPP measurements. After the UPP measurement has been performed, which is expected to take less than five minutes, general anaesthesia will then be changed to a level sufficient for the planned urological procedure.

Overactive sphincter These patients have presented to the bladder service with problems because of abnormality of sphincter activity. These children will be expected to have high tone sphincters. They may have varieties of diagnoses which include high tone non-relaxing sphincter, Fowler's syndrome and dysfunctional voiding. They will commonly have voiding symptoms such as hesitancy, straining, poor stream or the sensation of incomplete emptying. There is, perhaps, surprisingly high incidence of storage symptoms such as frequency urgency and incontinence.

A diagnosis of dysfunctional voiding will have been made based on voiding pelvic EMGs based on representative at least two representative voids.

The children to be recruited will require VCMG urodynamics as part of their clinical care. Patients who are recruited to this arm of the study will in addition have a urethral pressure profile measurement performed on the same day as their VCMG.

VCMG requires the insertion of urethral and rectal catheters. This is an invasive procedure. In a small group of children this is straightforward; these children perform intermittent catheterisation regularly to empty their bladder and so are used to having a catheter passed. However, in the majority passing a urethral catheter can be distressing and so in the investiators' unit catheter insertion for urodynamics is done either under general anaesthesia, for those under seven years, or with inhalational sedation (Entonox) for those above the age of seven years.

Subjects who participate in this arm of the study will undergo VCMG. The UPP measurement will be done immediately before the insertion of the bladder catheter. If sedation or anaesthesia is required for the catheter insertion this will have been administered, lignocaine gel will be applied to the urethra (standard for catheter insertion prior to VCMG), a UPP measurement taken, and then the catheters inserted for urodynamics.

Underactive sphincter Underactive sphincter results in the symptom of stress incontinence. In children the most common cause of urethral sphincter weakness is neurological disease that causes neuropathic bladder. These neurological conditions include children with spina bifida (e.g. myelomeningocele or closed spinal dysraphism). In the investigators' unit children with neuropathic bladder are frequently managed with intermittent catheterisation to empty their bladders and antimuscarinic medication to reduce bladder storage pressures; they undergo annual surveillance of their bladder with videocystometry urodynamics. They are familiar with catheters and VCMG.

Stress incontinence is an unusual symptom in children. In the investigators' unit these children are frequently investigated with VCMG.

Subjects recruited to this arm will either have symptoms of stress incontinence or have a neuropathic bladder associated with symptoms of urinary incontinence.

Subjects who participate in this arm of the study will undergo VCMG. The UPP measurement will be done immediately before the insertion of the bladder catheter. If sedation or anaesthesia is required for the catheter insertion this will have been administered, lignocaine gel will be applied to the urethra (standard for catheter insertion prior to VCMG), a UPP measurement taken, and then the catheters inserted for urodynamics.

The UPP's of these patients will be included for analysis if their subsequent urodynamics demonstrate either stress incontinence or continuous incontinence in the absence of simultaneous detrusor overactivity

Hypothesis:

Values and characteristics of MUCP during UPP measurement will be compared between the three groups to identify whether the groups can be distinguished based on these results. The hypothesis is that there are cut-off values for MUCP that can distinguish normal controls from those with overactive sphincter and also those with underactive sphincters.

ELIGIBILITY:
Inclusion Criteria All subjects • Age 7-16 years inclusive

Controls

* Concurrent urological disease requiring surgery which includes cystoscopy
* No significant urinary symptoms
* No day-time urinary incontinence
* Urinary frequency 4-7 per day
* No history of recurrent urinary infections (more than two infections in previous year)
* Has not passed a renal tract stone

Overactive sphincter

* Require VCMG as part of their clinical care
* A prior diagnosis of dysfunctional voiding. This will have been made in a neurologically intact child following previous non-invasive bladder investigation including two representative urine flows that demonstrate the following (Austin et al., 2014):

  * Intermittent and/or fluctuating flow rate
  * Pelvic EMG activity during voiding
* either perform intermittent catheterisation or have no contraindication to Entonox sedation (see below)

Underactive sphincter

* Have either:

  * Symptoms of stress urinary incontinence
  * Or urinary incontinence with a neuropathic bladder
* Require VCMG as part of their clinical care.
* either perform intermittent catheterisation or have no contraindication to Entonox sedation (see below)
* For the UPP data to be included for analysis their videocystometry should demonstrate o Stress urinary incontinence: defined as involuntary leakage of urine during increased abdominal pressure, in the absence of a detrusor contraction (Austin et al., 2014)

Exclusion Criteria:

* Unaccompanied by adult with parental responsibility who can give consent
* Previous bladder outlet or urethral surgery
* Other urological disease not mentioned specifically in the treatment group inclusion criteria; including posterior urethral valves, cerebral palsy, inherited metabolic disease
* Contraindication to Entonox if sedation required for catheter insertion:

  * Conditions where gas may be trapped in a body cavity, eg middle ear occlusion, intestinal obstruction
  * Unable to understand instruction for use of Entonox
* Evidence urinary tract infection on day UPP measurement

  * Symptoms of dysuria
  * Abnormally cloudy or offensive urine
  * Temperature of 38oc or more
* Urine dipstick positive nitrates or leucocytes on the day of the study, in the absence of a renal tract stone or indwelling catheter

Ages: 7 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Patients attending paediatric urology or bladder clinic
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
maximum urethral closure pressure (MUCP). | approximately 3 months
  Urodynamics finding

SECONDARY OUTCOMES:
Urethral pressure profile pattern | approximately 3 months
  Urodynamics finding

CONTACTS AND LOCATIONS:
Overall Officials: arash taghizadeh, mbbs, Principal Investigator — Evelina London Children's Hospital
Locations (1):
- Evelina London Children's Hosital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
there is no plan to share IPD

REFERENCES:
- [Background] Afshar K, Mirbagheri A, Scott H, MacNeily AE. Development of a symptom score for dysfunctional elimination syndrome. J Urol. 2009 Oct;182(4 Suppl):1939-43. doi: 10.1016/j.juro.2009.03.009. Epub 2009 Aug 20. PMID 19695637
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Vande Walle J, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J Urol. 2014 Jun;191(6):1863-1865.e13. doi: 10.1016/j.juro.2014.01.110. Epub 2014 Feb 4. PMID 24508614
- [Background] Bauer SB, Nijman RJ, Drzewiecki BA, Sillen U, Hoebeke P; International Children's Continence Society Standardization Subcommittee. International Children's Continence Society standardization report on urodynamic studies of the lower urinary tract in children. Neurourol Urodyn. 2015 Sep;34(7):640-7. doi: 10.1002/nau.22783. Epub 2015 May 21. PMID 25998310
- [Background] Comiter CV, Sullivan MP, Yalla SV. Correlation among maximal urethral closure pressure, retrograde leak point pressure, and abdominal leak point pressure in men with postprostatectomy stress incontinence. Urology. 2003 Jul;62(1):75-8. doi: 10.1016/s0090-4295(03)00123-7. PMID 12837426
- [Background] Dave S, Salle JL. Current status of bladder neck reconstruction. Curr Opin Urol. 2008 Jul;18(4):419-24. doi: 10.1097/MOU.0b013e328302edd5. PMID 18520766
- [Background] DeLancey JO, Trowbridge ER, Miller JM, Morgan DM, Guire K, Fenner DE, Weadock WJ, Ashton-Miller JA. Stress urinary incontinence: relative importance of urethral support and urethral closure pressure. J Urol. 2008 Jun;179(6):2286-90; discussion 2290. doi: 10.1016/j.juro.2008.01.098. Epub 2008 Apr 18. PMID 18423707
- [Background] Edwards L, Malvern J. The urethral pressure profile: theoretical considerations and clinical application. Br J Urol. 1974 Jun;46(3):325-35. doi: 10.1111/j.1464-410x.1974.tb03834.x. No abstract available. PMID 4858680
- [Background] Farhat W, Bagli DJ, Capolicchio G, O'Reilly S, Merguerian PA, Khoury A, McLorie GA. The dysfunctional voiding scoring system: quantitative standardization of dysfunctional voiding symptoms in children. J Urol. 2000 Sep;164(3 Pt 2):1011-5. doi: 10.1097/00005392-200009020-00023. PMID 10958730
- [Background] Fowler CJ, Kirby RS, Harrison MJ. Decelerating burst and complex repetitive discharges in the striated muscle of the urethral sphincter, associated with urinary retention in women. J Neurol Neurosurg Psychiatry. 1985 Oct;48(10):1004-9. doi: 10.1136/jnnp.48.10.1004. PMID 4056803
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Heron J, Grzeda MT, von Gontard A, Wright A, Joinson C. Trajectories of urinary incontinence in childhood and bladder and bowel symptoms in adolescence: prospective cohort study. BMJ Open. 2017 Mar 14;7(3):e014238. doi: 10.1136/bmjopen-2016-014238. PMID 28292756
- [Background] Jiang R, Kelly MS, Routh JC. Assessment of pediatric bowel and bladder dysfunction: a critical appraisal of the literature. J Pediatr Urol. 2018 Dec;14(6):494-501. doi: 10.1016/j.jpurol.2018.08.010. Epub 2018 Aug 28. PMID 30297226
- [Background] Meunier P, Mollard P. Urethral pressure profile in children: a comparison between perfused catheters and micro-transducers, and a study of the usefulness of urethral pressure profile measurements in children. J Urol. 1978 Aug;120(2):207-10. doi: 10.1016/s0022-5347(17)57110-4. PMID 671637
- [Background] Sihra N, Malde S, Panicker J, Kightley R, Solomon E, Hamid R, Ockrim J, Greenwell TJ, Pakzad M. Does the appearance of the urethral pressure profile trace correlate with the sphincter EMG findings in women with voiding dysfunction? Neurourol Urodyn. 2018 Feb;37(2):751-757. doi: 10.1002/nau.23341. Epub 2017 Jul 5. PMID 28678412
- [Background] Tran K, Kuo B, Zibaitis A, Bhattacharya S, Cote C, Belkind-Gerson J. Effect of propofol on anal sphincter pressure during anorectal manometry. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):495-7. doi: 10.1097/MPG.0000000000000190. PMID 24121151
- [Background] Wiseman OJ, Swinn MJ, Brady CM, Fowler CJ. Maximum urethral closure pressure and sphincter volume in women with urinary retention. J Urol. 2002 Mar;167(3):1348-51; discussion 1351-2. doi: 10.1016/s0022-5347(05)65297-4. PMID 11832729